CLINICAL TRIAL: NCT00036816
Title: Randomized Phase III Study Of Adjuvant Immunization With The NA17.A2 And Melanoma Differentiation Peptites In HLA-A2 Patients With Primary Ocular Melanoma At High Risk Of Relapse
Brief Title: Vaccine Therapy in Treating Patients With Melanoma of the Eye
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-18001 -88001; EORTC-18001; EORTC-88001
Record Dates: First submitted 2002-05-13; First posted 2003-01-27 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Intraocular Melanoma
Keywords: ciliary body and choroid melanoma, medium/large size
MeSH Terms: conditions — Uveal Melanoma | interventions — MART-1 Antigen

INTERVENTIONS:
Biological: MART-1 antigen
Biological: NA17-A antigen
Biological: gp100 antigen
Biological: tyrosinase peptide

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells and decrease the recurrence of melanoma of the eye.

PURPOSE: Randomized phase III trial to determine the effectiveness of vaccine therapy in treating patients who are at high risk for recurrent melanoma of the eye.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether adjuvant NA17-A and melanoma differentiation peptides are effective in decreasing the occurrence of liver metastasis in HLA-A2-positive patients with primary ocular melanoma at high risk of relapse.
* Determine whether this regimen increases survival of these patients.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to tumor size (medium vs large), prior treatment of primary tumor (surgery vs radiotherapy), and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive vaccination with NA17-A and melanoma differentiation peptides (e.g., tyrosinase, Melan-A, and gp100 antigens) subcutaneously and intradermally on days 1, 8, 15, and 22. Patients then receive a vaccination once every 14 days for 4 doses, once every 28 days for 4 doses, once every 56 days for 4 doses, and then once every 3 months for a total of 4 years.
* Arm II: Patients undergo observation only every 3 months for 2 years and then every 6 months for 2 years.

All patients are followed every 3 months for 1 year and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 600 patients (300 per treatment arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of ocular melanoma

  * No melanoma of the iris
* Disease adequately treated by prior surgery (enucleation or tumorectomy) and/or radiotherapy

  * No more than 5 weeks since the beginning of primary tumor treatment
* Measurable disease

  * At least 12.0 mm in largest diameter OR
  * At least 6.0 mm in height
* HLA-A2 positive
* No distant metastases

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Hemoglobin at least 9 g/dL
* Neutrophil count at least 2,000/mm^3
* Lymphocyte count at least 700/mm^3
* Platelet count at least 100,000/mm^3
* No bleeding disorder

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* AST and ALT no greater than 2 times upper limit of normal (ULN)
* Lactate dehydrogenase no greater than 2 times ULN
* Alkaline phosphatase no greater than 2 times ULN
* Gamma glutamyl transpeptidases no greater than 2 times ULN
* Hepatitis C antibody negative
* Hepatitis B antigen negative

Renal:

* Creatinine no greater than 2.0 mg/dL

Immunologic:

* No clinical immunodeficiency
* No autoimmune diseases
* No inflammatory bowel disease
* No active infection requiring antibiotics
* No multiple sclerosis

Other:

* HIV negative
* No other malignancy except surgically cured carcinoma in situ of the cervix or basal cell or squamous cell carcinoma of the skin
* No other uncontrolled illness
* No psychological, familial, sociological, or geographical conditions that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No other concurrent immunotherapy or biologic therapy

Chemotherapy:

* No concurrent chemotherapy

Endocrine therapy:

* At least 3 weeks since prior steroids
* No concurrent chronic therapy with high doses of corticosteroids (e.g., methylprednisolone at least 12 mg/day)
* Concurrent topical or inhalation steroids allowed
* No concurrent hormonal therapy

Radiotherapy:

* See Disease Characteristics
* Prior proton beam therapy allowed
* Prior brachytherapy without tumor resection allowed
* Recovered from prior radiotherapy
* No prior radiotherapy to the spleen
* No prior pre-enucleation radiotherapy
* No prior ruthenium Ru 106 as primary therapy alone
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* Prior transcleral tumor resection allowed
* Recovered from prior surgery
* No prior major organ allograft
* No prior splenectomy

Other:

* No other concurrent investigational drugs
* No concurrent systemic immunosuppressive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2002-02; Primary Completion 2003-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Brichard, MD, Study Chair — Cliniques universitaires Saint-Luc- Université Catholique de Louvain; Jan U. Prause, MD, Study Chair — University of Copenhagen
Locations (2):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- University of Copenhagen, Copenhagen, Denmark